CLINICAL TRIAL: NCT06328647
Title: Quantra Point-of-Care Hemostasis Monitoring and Perioperative Blood and Blood Component Transfusion During High-Risk Complex Cardiac Surgery: A Randomized Clinical Trial
Brief Title: Quantra Point-of-Care Hemostasis Monitoring
Acronym: QUANTRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-010
Record Dates: First submitted 2024-03-08; First posted 2024-03-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Bleeding; Hemostatic Disorder
MeSH Terms: conditions — Hemorrhage; Hemostatic Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and outcome assessor will be masked to the group allocation. Clinicians will be unmasked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- POC Quantra QPlus System (Experimental): Perfusion team or trained (certified for POC testing) research personnel will perform hemostasis testing using the Quantra QPlus POC System, results will be interpreted by the primary anesthesia team that will decide if transfusion of blood components is necessary in the operating room and up to 12 hours after surgery in the cardiac surgery intensive care unit (ICU).
  Interventions: Device: POC Quantra QPlus System
- Routine Care (Active Comparator): The primary anesthesia provider will determine the need for blood and blood component transfusion with or without guidance from central laboratory testing for hemostatic abnormalities in the operating room and up to 12 hours after surgery in the cardiac surgery intensive care unit (ICU).
  Interventions: Other: Routine care

INTERVENTIONS:
Device: POC Quantra QPlus System — The POC Quantra QPlus System will be located in the operating room. Samples will be processed by trained (certified for POC testing) personnel and interpreted by the primary anesthesia team. The anesthesia team will perform a baseline hemostatic assessment , approximately 15 min prior to separation from CPB, and again 10-20 min following protamine administration using the Quantra POC hemostasis monitor. If persistent bleeding occurs despite clinical management, coagulation will be rechecked by a repeated Quantra assessment and treated as necessary. A Quantra device will be placed in the ICU for assessment for the first 6 hours following surgery.
  Arms: POC Quantra QPlus System
Other: Routine care — Blood and blood component transfusions will be determined by provider preference based on clinical findings. The anesthesia caregiver will perform laboratory testing for coagulation management at his/her discretion. Usual laboratory testing may include assessment of TEG with heparinase, platelet count, fibrinogen concentration at approximately 30-40 min prior to separation from cardiopulmonary bypass. Another set of laboratory tests may be sent post-CPB including TEG, platelet count, fibrinogen concentration, PT/aPTT, INR. Anesthesia caregiver will treat clinical bleeding and coagulopathy at his/her discretion.
  Arms: Routine Care

SUMMARY:
The investigators will test the hypothesis that utilization of a blood and blood component transfusion algorithm guided by the POC Quantra QPlus System in patients undergoing complex cardiac surgery will reduce RBC, plasma, cryoprecipitate, and platelet transfusion during surgery and the first 12 postoperative hours, compared to standard of care (central laboratory transfusion monitoring at the primary anesthesia provider's discretion).

DETAILED DESCRIPTION:
The Investigators propose a randomized control trial to assess patients scheduled for aortic surgery or high-risk cardiac surgery requiring cardiopulmonary bypass.

Patients will be randomized 1:1 to routine care or POC Quantra QPlus System. The total number of blood and blood component transfusions (including RBC, plasma, cryoprecipitate, and platelets) during and after cardiac surgery until 12 hours after ICU arrival will be analyzed between the groups.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or more
2. Scheduled for aortic surgery or high-risk cardiac surgery requiring cardiopulmonary bypass (high-risk surgery includes reoperative surgery, active endocarditis, expected need for intraoperative circulatory arrest, radiation heart disease, end-stage kidney disease requiring renal replacement therapy, combination surgery including more than one valve or valve plus CABG, low left ventricular ejection fraction [EF<30%] with potential need for mechanical circulatory support with intra-aortic balloon pump, extracorporeal membrane oxygenation [ECMO], pulmonary thromboembolectomy or percutaneous left ventricular assist device (VAD), and planned placement of a durable left VAD with or without placement of RV assist device.

Exclusion Criteria:

1. Preoperative diagnosis of a pre-existing coagulation or bleeding disorder
2. Preoperative abnormal coagulation disorder (platelet count below 100,000/uL and/or aPTT >40 seconds in the absence of heparin therapy. Prolonged aPTT >40 seconds in the acceptable if due to heparin therapy.)
3. Liver disease, defined as a history of cirrhosis, liver enzymes >3x normal range or manifested by elevated PT suggesting abnormal liver synthetic function not explained by other comorbidities
4. Pregnancy or breastfeeding
5. Refusal to accept red blood cells and blood component transfusions.
6. Contraindications to proposed interventions.
7. Unable to understand English as a first language or unable comprehend the study and/or the consent forms.
8. Vulnerable patients including prisoners, human fetuses, and neonates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood and blood component transfusions | 12 hours after ICU arrival
  The total number of blood and blood component transfusions (including RBC, plasma, cryoprecipitate, and platelets) during and after cardiac surgery until 12 hours after ICU arrival.

SECONDARY OUTCOMES:
Bleeding | During hospitalization, up to 24 hours
  Postoperative bleeding assessed by the Universal Definition of perioperative bleeding during index hospitalization, which classification into categories 0 - 4 based upon the following complications related to perioperative bleeding: the assessment of delayed sternal closure; amount of postoperative chest tube blood loss within 12 hours; Units of PRBC, FFP, platelets, and cryoprecipitate; need for PCCs or rFVIIa, or re-exploration/tamponade.

OTHER OUTCOMES:
PT/aPTT | 1 Hour after surgery end
  Postoperative PT/aPTT measurement at 1 hour (±1 hr) after surgery end.
INR | 1 hour after surgery end
  Postoperative INR measurement at 1 hour (±1 hr) after surgery end.
Platelet | 1 hour after surgery end
  Postoperative platelet count measurement at 1 hour (±1 hr) after surgery end.
Fibrinogen | 1 hour after surgery end
  Postoperative fibrinogen measurement at 1 hour (±1 hr) after surgery end.
hematocrit/hemoglobin | 1 hour after surgery end
  Postoperative hematocrit/hemoglobin measured at 1 hour (±1 hr) after surgery end.
ICU length of stay | During hospitalization, an average of 30 days.
  ICU length of stay
Hospital length of stay. | During hospitalization, an average of 30 days.
  Hospital length of stay.
In-hospital mortality | During hospitalization
  In-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Andra Duncan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States